CLINICAL TRIAL: NCT03482427
Title: Assessing the Healthy Heart Score Intervention In the Primary Care Setting as a Primordial Prevention Tool
Brief Title: Healthy Heart Score Intervention In the Primary Care Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio University (Other)
Collaborators: OhioHealth (Other)
Responsible Party: Principal Investigator, Mercedes Sotos Prieto, PhD, Assistant Professor, Ohio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-X-35
Record Dates: First submitted 2018-03-13; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: We will test our intervention compared to usual care (control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): After completion of the Healthy Hear Score assessment, participants will receive a lifestyle intervention based on the Healthy Heart Score results for 12-weeks by trained dietetic interns on-site. Participants will receive a check-in email or phone 6 weeks after the initial visit. A Registered Dietitian is also available to speak with patients. The intervention will consist on educational materials based on each component of the Healthy Heart Score and other lifestyle behaviors
  Interventions: Behavioral: Healthy Heart Score
- Control (No Intervention): Participants in the control group will follow their usual care protocol after taking the Healthy Heart Score assessment. Researchers will provide the Healthy Heart Score survey results, but will not discuss or interpret the results with them. Participants can discuss any concern they have with their usual physician if they choose. After the follow-up visit and upon completion of the study, all participants in the control group may also receive the educational handouts and will be granted access to the Healthy Heart Score application if they wish.

INTERVENTIONS:
Behavioral: Healthy Heart Score — Educational materials based on each component of the Healthy Heart Score and other lifestyle behaviors will be provided to the participants that include the following topics: Fruit and vegetable consumption, Whole grain consumption/ limiting refined grains, Healthy protein choices, Healthy dietary fats, Limiting Sugar-sweetened beverages, Importance of physical activity, Proper hydration, Stress management, Adequate Sleep, Smoking Cessation, Weekly menu example, Recipe Cards following the Mediterranean diet principals, Interactive weekly checklist to encourage participants to meet their weekly goals for consumption of fruits, vegetable, nuts and seeds. Participants will receive a check-in email or phone 6 weeks after the baseline visit. A Registered Dietitian is also available to speak with patients.
  Arms: Intervention

SUMMARY:
In this pilot study, the investigators will assess the clinical utility and feasibility of the Healthy Heart Score in the primary clinical care setting for the primordial prevention of cardiovascular disease. The investigators will conduct a randomized clinical trial to test the lifestyle intervention based on the Healthy Heart Score compared to usual care. The aim is to include 100 participants (50 in each group). Each participant will complete 2 visits (initial and a follow up visit after 12 weeks).

DETAILED DESCRIPTION:
Created by the Harvard T.H Chan School of Public Health, the Healthy Heart Score is a previously validated online risk calculator that determines the 20-year Cardiovascular Disease ) risk based on 9 modifiable lifestyle factors including; smoking habits, body mass index, physical activity, alcohol consumption, fruit and vegetables intake, cereal fiber, nuts, sugar-sweetened beverages, and red meat, and processed meats consumption.

In this pilot study, the investigators will assess the clinical utility and feasibility of the Healthy Heart Score in the primary clinical care setting for the primordial prevention of cardiovascular disease. The investigators will conduct a clinical trial to test our intervention compared to usual care. The investigators will conduct a randomized clinical trial to test the lifestyle intervention based on the Healthy Heart Score compared to usual care. The aim is to include 100 participants (50 in each group). Each participant will complete 2 visits (initial and a follow up visit after 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, No cardiovascular diagnosis, Body Mass Index > 25 and/or having at least one of the following clinical risk factors: elevated blood pressure, pre-high cholesterol, pre-diabetes but not currently taking medications for the previous conditions.

Exclusion Criteria:

* Those not meeting the inclusion criteria and women who are pregnant or planning to get pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the overall Healthy Heart Score risk score | 12-weeks
  The Healthy Heart Score is a lifestyle-based risk tool that estimates 20-year CVD risk (https://healthyheartscore.sph.harvard.edu/) This gender-specific algorithm has been published (DOI: 10.1161/JAHA.114.000954):
  20-year CVD risk (%) "Healthy Heart Score" = [1 - 0. 9660 (exp [W- 6.57301)] × 100%
  where W= 0.10820 x age + 0.15285 (if past smoker) + 0.90138 (if current smoker) + 0.04676 × BMI - 0.01923 × grams/d of alcohol + 0.0004 × (grams/d of alcohol)2- 0.029251 × hours/week of physical activity - 0.05113 × diet score* 20-year CVD risk (%) "Healthy Heart Score" = [1 - 0. 96368 (exp [W-7.2437)] × 100%
  where W= 0.13580 x age- 0.0005 x (age)2 + 0.06979 (if past smoker) + 0.42305 (if current smoker) +0.07424 × BMI - 0.00898 × grams/d of alcohol + 0.0001 × (grams/d of alcohol)2- 0.01755 × hours/week of physical activity - 0.06691 × diet score
Changes in the overall composite of diet | 12-weeks
  women: Diet score = (0.03626 × grams/d of cereal fiber + 0.18283 [if fruits + vegetables ≥3 servings/d] + 0.14522 [if nuts 0.1-1 servings/d + 0.2444 [if nuts >1 servings/d]- 0.14631 × servings/d of sugar-sweetened beverages - 0.15624 × servings/d of red and processed meats)*10
  Women:
  Diet score = (0.03626 × grams/d of cereal fiber + 0.18283 [if fruits + vegetables ≥3 servings/d] + 0.14522 [if nuts 0.1-1 servings/d + 0.2444 [if nuts >1 servings/d]- 0.14631 × servings/d of sugar-sweetened beverages - 0.15624 × servings/d of red and processed meats)*10.
  Men:
  where W= 0.13580 x age- 0.0005 x (age)2 + 0.06979 (if past smoker) + 0.42305 (if current smoker) +0.07424 × BMI - 0.00898 × grams/d of alcohol + 0.0001 × (grams/d of alcohol)2- 0.01755 × hours/week of physical activity - 0.06691 × diet score*
Changes in fruit and vegetables intake | 12-weeks
  servings/day
Changes in red and processed meats intake | 12-weeks
  servings/week
Changes in sugar and sweetened beverages | 12-weeks
  servings/week
Changes in nut consumption | 12-weeks
  servings week
changes in alcohol consumption | 12-weeks
  g/day
changes in cereal fiber | 12-weeks
  g/day
changes in body mass index | 12-weeks
  kg/m2
Changes in physical activity | 12-weeks
  hours per week

SECONDARY OUTCOMES:
Changes in total cholesterol levels | 12-weeks
Changes in triglycerides levels | 12-weeks
Changes in Low Density Protein levels | 12-weeks
Changes in High Density Protein levels | 12-weeks
Changes in Hemoglobin glycosylated levels | 12- weeks
Changes in systolic blood pressure | 12-weeks
  mmHg
Changes in diastolic blood pressure | 12-weeks
  mmHg
changes in percentage of body fat | 12-weeks
changes in body weight | 12-weeks
  pounds/kg

CONTACTS AND LOCATIONS:
Overall Officials: Mercedes Sotos Prieto, PhD, Principal Investigator — Ohio University
Locations (1):
- OhioHealth Dublin Methodist Hospital, Dublin, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided